CLINICAL TRIAL: NCT07154875
Title: Randomized Controlled Trial of Assisted Hatching Timing (Day-3 vs Day-5) and Its Impact on Blastocyst Morphology and Genetic Outcomes in IVF Cycles Undergoing PGT-A
Brief Title: Day-3 vs Day-5 Assisted Hatching: Impact on Blastocyst Morphology and PGT-A Outcomes
Acronym: AH-PGTA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hoang Minh Ngan (Other)
Collaborators: 16A Ha Dong General Hospital (Other)
Responsible Party: Sponsor-Investigator, Hoang Minh Ngan, Principal Investigator, Embryologist, Head of IVF Laboratory, 16A Ha Dong General Hospital
Organization: 16A Ha Dong General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AH-PGTA-2025; 16A-IRB-2025 (Other: Institutional Review Board of 16A Ha Dong General Hospital)
Record Dates: First submitted 2025-08-27; First posted 2025-09-04 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Infertility; In Vitro Fertilization; Embryo Development
Keywords: Assisted hatching, Day-3 vs Day-5, Blastocyst morphology, Trophectoderm biopsy, PGT-A, Aneuploidy, Mosaicism
MeSH Terms: conditions — Infertility; Aneuploidy

STUDY DESIGN:
Intervention Model Description: Embryos randomized to receive assisted hatching on Day-3 (Arm A) or Day-5 (Arm B) prior to trophectoderm biopsy.
Who Masked: Outcomes Assessor
Masking Description: The PGT-A analysts evaluating the NGS results were blinded to the assisted hatching timing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Day-3 Assisted Hatching (Experimental): Embryos undergo laser-assisted zona drilling on Day-3. Embryos are then cultured to Day-5 and biopsied for PGT-A.
  Interventions: Procedure: Assisted Hatching
- Day-5 Assisted Hatching (Experimental): Embryos are cultured without zona drilling until Day-5. Laser-assisted hatching is performed immediately before trophectoderm biopsy for PGT-A.
  Interventions: Procedure: Assisted Hatching

INTERVENTIONS:
Procedure: Assisted Hatching — Laser-assisted zona drilling performed either on Day-3 or Day-5 of culture, depending on randomization arm.
  Other Names: Laser-assisted hatching; LAH; Zona drilling; AH

SUMMARY:
This randomized controlled trial evaluates the effect of assisted hatching (AH) timing on embryo development and genetic outcomes in in vitro fertilization (IVF) cycles with preimplantation genetic testing for aneuploidy (PGT-A). Eligible patients undergoing IVF with PGT-A will have embryos randomized to receive assisted hatching either on Day-3 or Day-5 of culture, prior to trophectoderm biopsy. The primary outcome is the rate of aneuploid blastocysts. Secondary outcomes include blastocyst morphology, expansion stage, and the correlation between morphology and genetic results. The study aims to determine whether earlier or later assisted hatching affects embryo viability and the accuracy of genetic testing. The trial will provide evidence to optimize laboratory protocols in IVF centers.

DETAILED DESCRIPTION:
This prospective randomized controlled trial compares two standardized laboratory procedures of assisted hatching (AH) timing in IVF cycles undergoing PGT-A. In Arm A, AH will be performed on Day-3 embryos; in Arm B, AH will be performed on Day-5 blastocysts prior to trophectoderm biopsy. A total of approximately 200 IVF cycles, involving around 650 embryos, will be included. Randomization will be conducted using block randomization. The primary outcome is the proportion of aneuploid blastocysts identified by next-generation sequencing (NGS). Secondary outcomes include blastocyst morphology (ICM, TE, expansion), biopsy efficiency, and correlation between morphological parameters and genetic outcomes.

All procedures are part of the routine IVF-PGT workflow, and no additional risks to patients are introduced beyond standard care. The trial has been approved by the Institutional Review Board of 16A Ha Dong General Hospital.

ELIGIBILITY:
Inclusion Criteria:

* IVF cycles with PGT-A
* Oocyte age 20-45 years (donor cycles: donor's age)
* AMH 1-10 ng/mL within 12 months
* AFC ≥5 follicles (2-9 mm, both ovaries, day 2-5)
* Controlled ovarian stimulation: antagonist or PPOS protocols
* Stratified analysis by age (<30, 30-34, 35-39, ≥40)
* Sperm source: ejaculated samples prepared by density-gradient or swim-up
* No surgical sperm retrieval
* No advanced sperm selection (IMSI, PICSI, MACS)

Exclusion Criteria:

* History of ≥3 failed IVF cycles or ≥3 consecutive miscarriages
* Indication for PGT-M or PGT-SR (monogenic disorders, translocations)
* Severe medical/autoimmune conditions affecting oocytes/embryos (e.g. uncontrolled diabetes, active lupus)
* No MII oocytes available for ICSI
* Embryos not eligible for biopsy per SOP (early zona hatching, degeneration, poor expansion)
* Sperm from surgical retrieval or advanced sperm selection (IMSI, PICSI, MACS)
* PCOS diagnosed by Rotterdam criteria (≥2/3 features)

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-06-14 (Actual); Primary Completion 2026-12-14 (Estimated); Study Completion 2028-06-14 (Estimated)

PRIMARY OUTCOMES:
Proportion of aneuploid blastocysts | At the time of trophectoderm biopsy and PGT-A result (Day 5-6 of embryo culture).
  Percentage of blastocysts diagnosed as aneuploid by next-generation sequencing (NGS) after trophectoderm biopsy in each group (Day-3 vs Day-5 AH).

SECONDARY OUTCOMES:
Blastocyst morphology (ICM and TE grade) | Day 5-6 of culture
  Comparison of blastocyst inner cell mass (ICM) and trophectoderm (TE) grading between Day-3 and Day-5 AH groups.
Mosaicism rate | Day 5-6 of culture
  Proportion of blastocysts diagnosed as mosaic by NGS in each group.

OTHER OUTCOMES:
Correlation between blastocyst morphology and genetic outcome | Day 5-6 of culture (at the time of trophectoderm biopsy and PGT-A result)
  Analysis of the correlation between blastocyst morphology (ICM and TE grade, expansion stage) and genetic outcomes (euploid, aneuploid, mosaic).

CONTACTS AND LOCATIONS:
Overall Officials: Ngan M Hoang, MSc, Principal Investigator — Center for Reproductive Support, 16A Ha Dong General Hospital; Tao D Nguyen, MD, PhD, Professor, Study Chair — Center for Reproductive Support, 16A Ha Dong General Hospital
Locations (1):
- Center for Reproductive Support, 16A Ha Dong General Hospital, Hanoi, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided
The plan for sharing individual participant data (IPD) has not been finalized. De-identified embryo-level data may be shared upon reasonable request for academic purposes after study completion.

REFERENCES:
- [Background] ESHRE Working Group on Recurrent Implantation Failure; Cimadomo D, de Los Santos MJ, Griesinger G, Lainas G, Le Clef N, McLernon DJ, Montjean D, Toth B, Vermeulen N, Macklon N. ESHRE good practice recommendations on recurrent implantation failure. Hum Reprod Open. 2023 Jun 15;2023(3):hoad023. doi: 10.1093/hropen/hoad023. eCollection 2023. PMID 37332387
- [Background] McArthur SJ, Leigh D, Marshall JT, de Boer KA, Jansen RP. Pregnancies and live births after trophectoderm biopsy and preimplantation genetic testing of human blastocysts. Fertil Steril. 2005 Dec;84(6):1628-36. doi: 10.1016/j.fertnstert.2005.05.063. PMID 16359956
- [Background] Capalbo A, Rienzi L, Cimadomo D, Maggiulli R, Elliott T, Wright G, Nagy ZP, Ubaldi FM. Correlation between standard blastocyst morphology, euploidy and implantation: an observational study in two centers involving 956 screened blastocysts. Hum Reprod. 2014 Jun;29(6):1173-81. doi: 10.1093/humrep/deu033. Epub 2014 Feb 26. PMID 24578475
- See also: Official website of 16A Ha Dong General Hospital - Center for Reproductive Support — https://benhvien16a.com/